CLINICAL TRIAL: NCT03372863
Title: Validation of Automated Ultrasound Method for Measurement of Cardiac Output: A Clinical Observational Study
Brief Title: Validation of Automated Cardiac Output Measurement
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 30112017
Record Dates: First submitted 2017-12-01; First posted 2017-12-14 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Output, Low; Surgery
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac surgery patients

SUMMARY:
Automated software analysis now allows for quick estimation of cardiac output from the echocardiographic 5-chamber view. This study will validate the automated software method against pulmonary artery thermodilution and against conventional cardiac output measurement with echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative cardiac surgery patient
* Pulmonary artery catheter in situ
* Extubated

Exclusion Criteria:

* No echocardiographic image available
* No consent
* Moderat-severe aortic insufficiency
* Moderat-severe tricuspid insufficiency
* Moderat-severe mitral valve insuffficiency
* Arythmia Intracardiac shunt Moderat-severe hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative cardiac surgery patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of cardiac output measurement | 10 minutes
  Mean bias with limits of agreement for cardiac output measurement between automated cardiac output measurement and pulmonary artery thermodilution

SECONDARY OUTCOMES:
Trending ability | 120 minutes
  Trending ability for cardiac output measurement for automated cardiac output measurement compared to pulmonary artery thermodilution
Accuracy of cardiac output measurement | 10 minutes
  Mean bias with limits of agreement for cardiac output measurement between automated cardiac output measurement and conventional echocardiographic cardiac output measurement
Trending ability | 120 minutes
  Trending ability for cardiac output measurement for automated cardiac output measurement compared to traditional echocardiographic cardiac output measurement
Accuracy of cardiac output measurement | 10 minutes
  Mean bias with limits of agreement for cardiac output measurement between traditional cardiac output measurement and pulmonary artery thermodilution
Trending ability | 120 minutes
  Trending ability for cardiac output measurement for traditional echocardiographic cardiac output compared to pulmonary artery thermodilution

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Juhl-Olsen P, Smith SH, Grejs AM, Jorgensen MRS, Bhavsar R, Vistisen ST. Automated echocardiography for measuring and tracking cardiac output after cardiac surgery: a validation study. J Clin Monit Comput. 2020 Oct;34(5):913-922. doi: 10.1007/s10877-019-00413-w. Epub 2019 Nov 1. PMID 31677135